CLINICAL TRIAL: NCT00331643
Title: Phase II Trial of Ixabepilone (BMS-247550), an Epothilone B Analog, in Children and Young Adults With Refractory Solid Tumors
Brief Title: Ixabepilone in Treating Young Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01826; NCI-2012-01826 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL0524; CDR0000472912; NCI-P6451; NCI-06-C-0146; ADVL0524 (Other: Children's Oncology Group); ADVL0524 (Other: CTEP); U10CA098543 (NIH); NCT00318526 (obsolete NCT alias)
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-01

CONDITIONS: Adult Rhabdomyosarcoma; Adult Synovial Sarcoma; Alveolar Childhood Rhabdomyosarcoma; Childhood Synovial Sarcoma; Embryonal Childhood Rhabdomyosarcoma; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Neuroblastoma; Recurrent Osteosarcoma; Recurrent Wilms Tumor and Other Childhood Kidney Tumors
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma, Synovial; Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Neuroblastoma; Osteosarcoma; Wilms Tumor | interventions — ixabepilone

ARMS (1):
- Treatment (ixabepilone) (Experimental): Patients receive ixabepilone IV over 1 hour on days 1-5. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: ixabepilone

INTERVENTIONS:
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra

SUMMARY:
This phase II trial is studying how well ixabepilone works in treating young patients with refractory solid tumors. Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate to ixabepilone in various strata of recurrent solid malignant tumors of childhood and young adulthood, including all of the following: Embryonal or alveolar rhabdomyosarcoma, osteosarcoma, Ewing's sarcoma/peripheral neuroectodermal tumor, synovial sarcoma or malignant peripheral nerve sheath tumor, Wilms' tumor, and neuroblastoma.

II. Determine the time to progression for each tumor stratum. III. Prospectively evaluate the feasibility and utility of automated volumetric tumor measurement in patients with measurable pulmonary metastases, and descriptively compare volumetric measurements to 1-dimensional (RECIST criteria) and 2-dimensional (WHO criteria) measurements.

IV. Define and describe the toxicities of ixabepilone.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (Ewing's sarcoma/ peripheral neuroectodermal tumor vs osteosarcoma vs alveolar or embryonal rhabdomyosarcoma vs Wilms' tumor vs neuroblastoma vs synovial sarcoma/malignant peripheral nerve sheath tumor).

Patients receive ixabepilone IV over 1 hour on days 1-5. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed up every year for 5 years.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis (at original diagnosis or recurrence) of 1 of the following:

  * Embryonal or alveolar rhabdomyosarcoma
  * Osteosarcoma*
  * Ewing's sarcoma /peripheral neuroectodermal tumor*
  * Synovial sarcoma or malignant peripheral nerve sheath tumor*
  * Wilms' tumor*

    * Age ≤ 21 years at original diagnosis
  * Neuroblastoma

    * Age ≤ 21 years at original diagnosis
    * Clinically or radiographically measurable or evaluable (by iodine I 123 metaiodobenzoguanine sulfate [^123I-MIBG] or bone scan [evaluable tumors must be positive at ≥ 1 site])

      * If lesion was previously irradiated, a biopsy must be performed ≥ 6 weeks after completion of radiotherapy and viable neuroblastoma must be demonstrated
      * No elevated urinary catecholamines and/or bone marrow evidence of tumor with measurable disease clinically or by imaging modalities (CT scan, MRI, ^123I-MIBG, or bone scan)
* Refractory or recurrent disease with no known curative treatment options
* ECOG performance status (PS) 0-2 OR Karnofsky PS 50-100% (patients > 16 years of age) OR Lansky PS 50-100% (patients ≤ 16 years)
* Life expectancy ≥ 8 weeks
* No evidence of active graft-versus-host disease
* Absolute neutrophil count ≥ 1,500/mm³ (no growth factors)
* Platelet count ≥ 75,000/mm³ (transfusion independent)
* Not pregnant or nursing
* Fertile patients must agree to use effective contraception
* Negative pregnancy test
* Hemoglobin ≥ 8 g/dL (may receive RBC transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2.5 times ULN
* No clinically significant unrelated systemic illness that would preclude study treatment, including any of the following:

  * Serious infections
  * Hepatic, renal, or other organ dysfunction
  * CNS toxicity ≤ grade 2
  * No pre-existing sensory or motor neuropathy ≥ grade 2
* Seizure disorder allowed provided it is well controlled by anticonvulsants
* No known prior severe hypersensitivity reaction to agents containing Cremophor EL®
* Fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy
* More than 2 weeks since prior myelosuppressive chemotherapy (4 weeks if prior nitrosourea)
* At least 7 days since prior biologic agents
* At least 2 weeks since prior local palliative (small-port) radiotherapy
* At least 6 months since prior craniospinal radiotherapy OR radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* At least 4 months since prior allogeneic stem cell transplant (SCT)
* At least 2 months since prior autologous SCT
* No prior taxane (paclitaxel, docetaxel) therapy
* More than 1 week since prior growth factor use (except epoetin alfa)
* More than 1 week since prior and no concurrent strong inhibitors ofCYP3A4, including any of the following:

  * Clarithromycin
  * Troleandomycin
  * Erythromycin
  * Ketoconazole
  * Itraconazole
  * Fluconazole (doses > 3mg/kg/day)
  * Voriconazole
  * Nefazodone
  * Fluvoxamine
  * Verapamil
  * Diltiazem
  * Amiodarone
  * Grapefruit juice
* More than 1 week since prior and no concurrent enzyme-inducing anticonvulsants, including any of the following:

  * Carbamazepine
  * Felbamate
  * Phenobarbital
  * Phenytoin
  * Primidone
  * Oxcarbazepine
* No concurrent aprepitant
* No concurrent Hypericum perforatum (St. John's wort)
* No concurrent sargramostim (GM-CSF) or interleukin-11
* No other concurrent chemotherapy or immunomodulating agents
* No concurrent radiotherapy
* Concurrent steroids allowed for pain or chemotherapy-associated nausea or vomiting

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2006-04; Primary Completion 2007-10 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Time to progression | From enrollment until disease progression, death because of treatment complications, resection of measurable tumor or last patient follow-up whichever is first, assessed up to 5 years
  Estimated using the product-limit method of Kaplan and Meier.
Progression-free survival (PFS) | At 6 months
  The probability of PFS at 6 months will be summarized.
Response rate (complete response [CR] and partial response [PR]) according to Response Evaluation Criteria in Solid Tumor (RECIST) and World Health Organization (WHO) criteria | Up to 5 years
  Response rates will be calculated as the percent of patients whose best response is a CR or PR, and the fraction of responses obtained will have a 95% confidence interval, which takes into consideration the two-stage nature of the design.
Toxicity as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 5 years
  Toxicity information recorded will include the type, severity, time of onset, time of resolution, and the probable association with the study regimen. Tables will be constructed to summarize the observed incidence by severity and type of toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Widemann, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States